CLINICAL TRIAL: NCT06963645
Title: Augmented Reality-based Telerehabilitation Platform for Patients With Stroke: A Feasibility Study
Brief Title: Augmented Reality-based Telerehabilitation Platform for Patients With Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Maarten Lansberg, Professor of Neurology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 80062
Record Dates: First submitted 2025-04-30; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Telerehabilitation Group (Experimental): Participants will use a mobile medical device in a augmented reality (AR) headset for 30 minutes daily to support their rehabilitation process after stroke by completing assessments and training programs.
  Interventions: Device: AR rehabilitation app

INTERVENTIONS:
Device: AR rehabilitation app — The intervention will consist of an 8-week home rehabilitation program during which the participant will have 1) a total of 7 weekly remote video visits with a therapist and 2) daily at-home exercises using the AR headset with rehabilitation app, done independently.
  Other Names: Reia

SUMMARY:
The study is to 1) determine the feasibility of the use of our augmented reality (AR) rehabilitation program, including its preliminary efficacy, 2) determine the feasibility of obtaining an augmented reality assessment based on the Fugl-Meyer Assessment - Upper Extremity (FMA-UE).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. ≥3 months post ischemic or hemorrhagic stroke
3. Upper extremity deficit with an FMA-UE score between 20-50
4. Able to operate the AR device independently or with the help of a caregiver
5. Sufficiently proficient in the English language to follow instructions from Reia

Exclusion Criteria:

1. History of developmental, neurological or psychological impairment leading to functional disability
2. Vision or visual field impairment that interferes with the use of the AR headset
3. Severe photosensitivity that makes use of the AR headset uncomfortable
4. History of visually provoked seizures
5. Hearing aids
6. Cardiac pacemaker
7. Implantable cardioverter-defibrillator (ICD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Adherence | 8 weeks
  Percentage of days during the 8-week intervention period that a patient completes their 30-minute rehabilitation session.
Percentage of participants who successfully complete the vFMA-UE | Day 70
  Feasibility of obtaining the Fugl-Meyer Assessment - Upper Extremity (vFMA-UE) unsupervised, described by the percentage of participants who successfully complete the vFMA-UE at home on day 70, among patients who attempted to do the unsupervised vFMA-UE.

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Lansberg, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No